CLINICAL TRIAL: NCT00532181
Title: A Randomized Control Trial of Micro-Health Insurance in Cambodia
Brief Title: Micro-Health Insurance in Cambodia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, Berkeley (Other)
Collaborators: French Development Agency (Other Government); United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CPHS Protocol 2007-3-48
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Health Insurance Sale; Health Utilization; Asset Sales, Investment and Saving Behaviors
Keywords: Health insurance; Health utilization rates; Saving Behavior; Risk aversion

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: Savings Behavior and Consumer's Approach to Risk

SUMMARY:
People who buy insurance are sicker and/or more risk averse than those who don't. Also, Micro-health insurance increases utilization of public health care facilities and protects against asset sales.

DETAILED DESCRIPTION:
Randomly assign coupons giving a discounted price for insurance. Since coupon receipt is exogenous, use these coupons as an instrument for take-up of insurance.

ELIGIBILITY:
Inclusion Criteria:

* Must be in a village where the health insurance program is being offered.

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2008-04; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Better Understand Health Utilization Behavior in Cambodia

SECONDARY OUTCOMES:
Better Understand asset sales, investment and saving behaviors

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, PhD Econ, Principal Investigator — University of California, Berkeley
Locations (1):
- Sky Health Insurance, Phenom Phen, Cambodia